CLINICAL TRIAL: NCT00836433
Title: CONNECT for Better Falls Prevention in VA Community Living Centers
Acronym: CONNECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: EDU 08-417
Record Dates: First submitted 2009-02-02; First posted 2009-02-04 (Estimated); Results first posted 2014-10-30 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2014-10

CONDITIONS: Accidental Falls
Keywords: staff education; complexity science; social constructivist theory

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FALLS only (Active Comparator): Traditional falls educational intervention, including self-study modules, audit and feedback, falls team training, academic detailing, and toolkit.
  Interventions: Behavioral: FALLS educational intervention
- CONNECT and FALLS (Experimental): CONNECT educational intervention is designed to improve relationship-building and communication. The intervention includes 2 in-class session, group mapping exercise, individual relationship mapping exercises, Self-monitoring of interactions, individual staff coaching sessions. FALLS is a traditional falls educational intervention, including self-study modules, audit and feedback, falls team training, academic detailing, and toolkit.
  Interventions: Behavioral: CONNECT educational intervention; Behavioral: FALLS educational intervention

INTERVENTIONS:
Behavioral: CONNECT educational intervention — The CONNECT educational intervention is a training program for staff to improve communication with a more dense network of co-workers, in order to improve resident problem-solving. Includes in class sessions, group and individual mapping exercises, self-monitoring of interactions, and individual staff coaching.
  Arms: CONNECT and FALLS
Behavioral: FALLS educational intervention — FALLS is a traditional falls quality improvement education program including online modules, audit and feedback, and academic detailing sessions

SUMMARY:
This is a randomized trial of 2 nursing home staff educational approaches to reduce falls in VA nursing home (CLC) residents. One is a traditional falls education program using web-based modules, feedback of quality indicators, and meetings with influential peers. The other is a 12 week program that trains staff to form better connections and use effective communication strategies with a diverse network of co-workers, so that problem solving about resident problems is enhanced. The study will test whether the second intervention increases the effectiveness of the traditional falls education program.

DETAILED DESCRIPTION:
Background:

The current standard to improve resident outcomes in VA nursing homes combines educational programs and quality improvement processes. These educational programs typically focus on individual staff members' behavior and mastery of content, and use such instructional techniques as didactic modules, audit and feedback of individual performance, and academic detailing by influential peers. However, social constructivism theory and complexity science suggests that learning is a social process that occurs within the context of the relationships and interactions of the individual in their environment. Thus, traditional QI educational programs will not result in optimal changes in staff behavior unless a context is present which allows social learning to occur.

Objectives:

Based on social constructivist theory, complexity science, and prior research we have developed an educational intervention (CONNECT) that teaches staff to improve connections within and between disciplines, improve information flow, and seek out cognitive diversity in problem-solving about resident issues. The objectives of this study are to: (a) determine whether CONNECT improves staff interaction measures, fall-related process measures, and fall rates when combined with standard training on fall risk factor reduction, and (b) use the insights gained about social constructivist learning in CLCs to develop other educational interventions that address multi-factorial geriatric syndromes and system issues such as patient safety in VA nursing homes.

Methods:

To achieve these objectives we are conducting a randomized, controlled, single-blind study in which nursing homes receive either CONNECT plus a falls QI educational intervention (FALLS) or FALLS alone. Four VA CLCs in VISN-6 will participate, with an estimated n=144 participating staff members, and n=340 unique individuals with falls. The CONNECT intervention will be delivered over 3 months, and includes interactive in-class learning sessions, unit-based mentoring, and relationship mapping, all focused on helping staff build networks and relationships for problem-solving. The FALLS intervention will be delivered over 3 months either alone or after the CONNECT intervention. It includes web-based modules, audit and feedback, and academic detailing, all focused on individual fall reduction behaviors. Measurement is performed prior to intervention (all measures), at the conclusion of intervention (staff interaction measures, work environment measures, and social constructivist learning focus groups), and 6 months after the intervention (fall-related process and outcome measures). Analysis will use mixed models to account for the complex nesting of patients and staff within facilities.

Status:

Funding will begin on August 1, 2009 with anticipated intervention start time of January, 2010.

ELIGIBILITY:
Inclusion Criteria:

* All clinical and support staff in participating VA Community Living Centers

Exclusion Criteria:

* Inability to speak and understand English

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 689 (Actual)
Dates: Start 2010-02; Primary Completion 2011-10 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathleen S. Colon-Emeric, MD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (4):
- United States (4):
  - VA Medical Center, Asheville, Asheville, North Carolina
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - VA Medical Center, Salem VA, Salem, Virginia

REFERENCES:
- [Result] Colon-Emeric CS, Lyles KW, Su G, Pieper CF, Magaziner JS, Adachi JD, Bucci-Rechtweg CM, Haentjens P, Boonen S; HORIZON Recurrent Fracture Trial. Clinical risk factors for recurrent fracture after hip fracture: a prospective study. Calcif Tissue Int. 2011 May;88(5):425-31. doi: 10.1007/s00223-011-9474-4. Epub 2011 Feb 18. PMID 21331567
- [Result] Anderson RA, Corazzini K, Porter K, Daily K, McDaniel RR Jr, Colon-Emeric C. CONNECT for quality: protocol of a cluster randomized controlled trial to improve fall prevention in nursing homes. Implement Sci. 2012 Feb 29;7:11. doi: 10.1186/1748-5908-7-11. PMID 22376375
- See also: Pubmed reference link — http://www.ncbi.nlm.nih.gov/pubmed/24279686
- See also: Pubmed reference link — http://www.ncbi.nlm.nih.gov/pubmed/23704219

RESULTS

PARTICIPANT FLOW:
Groups:
- FALLS Only: Traditional falls educational intervention
  FALLS educational intervention: Traditional falls quality improvement education program including online modules, audit and feedback, and academic detailing sessions
- CONNECT + FALLS: CONNECT intervention on relationship-building and communication
  CONNECT educational intervention: Training program for staff to improve communication with a more dense network of co-workers, in order to improve resident problem-solving
  FALLS educational intervention: Traditional falls quality improvement education program including online modules, audit and feedback, and academic detailing sessions
Period: Overall Study
Arm/Group | FALLS Only | CONNECT + FALLS
Started | 361 | 328
Completed | 349 | 321
Not Completed | 12 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FALLS Only | CONNECT + FALLS | Total
Number analyzed (Participants) | 361 | 328 | 689
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (6) | 42 (5) | 44 (5)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 361 | 328 | 689
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 307 | 285 | 592
  Male | 54 | 43 | 97
Region of Enrollment [Number; unit: participants]
  United States | 361 | 328 | 689

OUTCOME MEASURES:

1. Primary Outcome: Fall-related Process Measures
Description: The proportion of applicable fall quality indicators documented for residents with falls during the study period. Quality indicators are specific fall risk assessment or prevention activities including orthostatic blood pressure assessment, vision assessment, environmental modification (bedroom, bathroom), footwear change, physical or occupational therapy referral, psychoactive medication reduction.
Time Frame: 6 months
Population: Note that the number of participants analyzed is not the same as the number of participants in the flow module. This is because this outcome measure is based not on the consented staff participants in the intervention, but resident charts abstracted in the pre and post intervention periods (waiver of consent obtained).
Measure: Mean (Standard Deviation); unit: proportion of indicators completed
Groups:
- FALLS: Traditional falls educational intervention
  FALLS educational intervention: Traditional falls quality improvement education program including online modules, audit and feedback, and academic detailing sessions
Arm/Group | FALLS | CONNECT + FALLS
Number analyzed (Participants) | 293 | 358
proportion of indicators completed | 0.40 (0.16) | 0.32 (0.13)

2. Secondary Outcome: Change in Facility Fall Rates
Description: Change in the risk-adjusted facility fall rates in the 6 months post intervention(s) compared to the 6 months before the intervention(s).
Time Frame: 6 months
Population: This is a facility level analysis of the fall rates in the 4 facilities randomized to FALLS alone compared to the 4 receiving CONNECT + FALLS. Within these groups, medical records from 293 and 358 residents with falls were abstracted to calculate the fall rates, therefore the "number of participants analyzed" is not the same as the flow module.
Measure: Number; unit: change in falls per bed per year
Units Other Than Participants: facilities
Groups:
- FALLS Only: Traditional falls educational intervention, including self-study modules, audit and feedback, falls team training, academic detailing, and toolkit.
  FALLS educational intervention: Traditional falls quality improvement education program including online modules, audit and feedback, and academic detailing sessions
- CONNECT and FALLS: CONNECT intervention on relationship-building and communication. Includes 2 in-class session, group mapping, individual relationship mapping, coaching sessions.
  CONNECT educational intervention: Training program for staff to improve communication with a more dense network of co-workers, in order to improve resident problem-solving
  FALLS educational intervention: Traditional falls quality improvement education program including online modules, audit and feedback, and academic detailing sessions
Arm/Group | FALLS Only | CONNECT and FALLS
Number analyzed (Participants) | 293 | 358
Number analyzed (facilities) | 4 | 4
change in falls per bed per year | 0.03 | -0.28

ADVERSE EVENTS:
Time Frame: 6 months
Description: During intervention delivery only
Arm/Group | FALLS Only | CONNECT + FALLS
Serious Adverse Events (participants affected / at risk) | 0/361 | 0/328
Other Adverse Events (participants affected / at risk) | 0/361 | 0/328

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No